CLINICAL TRIAL: NCT06719531
Title: SYNERGY PLUS: Evaluation of Next Generation Sensors (NGS) and Algorithm in Patients With Type 1 and Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The device is no longer under development.
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP345
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects with diabetes wearing DS5 (Experimental): Subjects wearing DS5 over 7-14 days and participating in FSTs
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — CGM and frequent sample testing

SUMMARY:
The purpose of this study is to find out how well a new continuous glucose monitor works for people with diabetes. This study will test the performance of the study sensor(s) for 7-14 days of wear in patients who are 11-80 years old with type 1 or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 11-80 years at time of screening.
2. Has a clinical diagnosis of type 1 or type 2 diabetes for 6 months or more, as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
3. Does not require a legally authorized representative to consent on their behalf due to mental or intellectual disability.
4. Subject or parent(s)/guardian(s) is/are literate and able to read the language offered in the study materials.
5. Subject and/or legally authorized representative is willing to provide informed consent for participation.
6. Has adequate venous access as assessed by investigator or appropriate staff.
7. Is willing to perform fingerstick blood glucose measurements as needed.
8. Is willing to wear the study devices continuously throughout the study.

Exclusion Criteria:

1. Has a history of 1 or more episodes of severe hypoglycemia during the 6 months prior to screening visit.
2. Has had a hypoglycemic seizure within the past 6 months prior to screening visit.
3. Has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to enrollment.
4. Has a history of allergy to dexamethasone or has been told by health care provider they may not take any products containing dexamethasone.
5. Has a history of 1 or more episodes of DKA in the last 6 months prior to screening visit.
6. Has a history of a seizure disorder.
7. Has a central nervous system or cardiac disorder resulting in syncope.
8. Will not tolerate tape adhesive in the area of sensor placement as assessed by a qualified individual.
9. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
10. Is pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD or implant).
11. Has diagnosis of adrenal insufficiency.
12. Is using hydroxyurea at time of screening or plans to use it during the study.
13. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks. (Please note participation in an observational study is acceptable.)
14. Has a planned procedure involving the use of a Magnetic Resonance Imaging (MRI), diathermy devices, or other devices that generate strong magnetic fields (e.g., x-ray, CT scan, or other types of radiation) during the study wear period.
15. Has elective surgery or hospitalization planned during the course of the study.
16. Has a clinical diagnosis of type 1 and is using pramlintide (Symlin), DPP-4 inhibitor, GLP-1 receptor agonist, metformin, and/or SGLT2 inhibitor at time of screening.
17. Is currently abusing illicit drug(s).
18. Is currently abusing marijuana.
19. Is currently abusing prescription medication(s).
20. Is currently abusing alcohol.
21. Has a hematocrit (Hct) more than 10% below the lower limit of normal reference range (please note that patients may use prior blood draw from routine care as long as done within 6 months of screening and report of lab placed with subject source documents).
22. Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances.
23. Has had any of the following cardiovascular events 1 year or more prior to screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances. Subject may be enrolled if clearance from a cardiologist is provided prior to or at screening.
24. Has any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
25. Is a member of the research staff involved with the study.
26. Is a Medtronic Diabetes employee or their immediate family member (excluding adult children and/or adult siblings).

Ages: 11 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints | The subject's participation from study enrollment to study exit is approximately 7 to 44 days.
  Descriptive summary will be used to characterize:
  • Skin assessment of subject's glucose sensor insertion sites

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - ProSciento, Chula Vista, California
  - John Muir Health, Concord, California
  - Headlands Research California, LLC, Escondido, California
  - Sansum Diabetes Research Institute, Goleta, California
  - Rady Children's Hospital, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Mills-Peninsula Medical Center: Diabetes Research Institute, San Mateo, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Atlanta Diabetes, Atlanta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Center, West Des Moines, Iowa
  - Barry J Reiner, MD, LLC, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Northwell Health, New Hyde Park, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - ClinRé 001-007, Bartlett, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Tekton Research, McKinney, Texas
  - Texas Diabetes & Endocrinology, Round Rock, Texas
  - Diabetes & Glandular Disease Clinic, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No